CLINICAL TRIAL: NCT04800978
Title: An Open Label, Single Arm, Safety Lead-in, Multicenter, Investigator Initiated Trial of Combination of Durvalumab , An Immune Checkpoint Inhibitor, and BVAC-C, A Cell-based Immunotherapeutic Vaccine, in Patients With HPV 16 or 18 Positive Cervical Cancer Failure to First-Line Platinum-based Chemotherapy
Brief Title: Combination of Durvalumab and BVAC-C in Patients With HPV 16 or 18 Positive Cervical Cancer Failure to First-Line Platinum-based Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-18-14325
Record Dates: First submitted 2021-01-11; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-01

CONDITIONS: Cervical Cancer
Keywords: BVAC-C; Durvalumab; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: •Part A: Open-labeled; 3+3 dose-escalation; Multi-center; safety lead-in phase
  •Part B: Open-labeled; Non-randomized, Single arm; Multi-center, efficacy evaluation phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BVAC-C+Durvalumab (Experimental): • Part A: The primary objective of the part A is to assess the maximum tolerable dose of BVAC-C combined with durvalumab 1500 mg as defined by dose-limiting toxicities (DLTs), and to find the maximum tolerated dose (MTD) that can be safely used for Part B (single arm phase II).
  • Part B: The primary objective of the part B is to evaluate the safety and clinical efficacy, as measured by 6-month PFS rate, of the combination therapy of durvalumab and BVAC-C in patients with HPV 16 or 18 positive cervical cancer recurrent after or refractory to first-line platinum-based chemotherapy +/-bevacizumab.
  Interventions: Biological: BAVC-C+Durvalumab

INTERVENTIONS:
Biological: BAVC-C+Durvalumab — * Durvalumab Durvalumab will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for infusion after dilution.
  * BVAC-C BVAC-C will be supplied in cyclic olefin co-polymer vials containing 1x10⁸ cells of suspension at a concentration of 5x10⁷ cells/mL infusion

SUMMARY:
This is an exploratory, open label, multi-center trial to evaluate the safety and efficacy of combination of durvalumab with BVAC-C in patients with cervical cancer refractory to or relapse after platinum-based first-line chemotherapy with safety lead-in phase.

The study consists of 2 parts: part A, a safety lead-in phase, and part B, an exploratory safety and efficacy evaluation phase.

Part A will be conducted as a 3+3 dose escalation manner, and part B will be conducted as a non-randomized single arm study.

•Part A: Open-labeled; 3+3 dose-escalation; Multi-center; safety lead-in phase

•Part B: Open-labeled; Non-randomized, Single arm; Multi-center, efficacy evaluation phase

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Willing and ability to provide blood and tumor tissue samples
* Histologically confirmed HPV 16/18-positive cervical carcinoma (squamous cell carcinoma; adenocarcinoma, adenosquamous carcinoma)
* Prior primary therapy with radical surgery, radical surgery followed by radiotherapy (+/- chemo), chemotherapy, or primary concurrent chemoradiotherapy
* Cervical cancer recurrent after or refractory to only 1 prior first-line platinum-based chemotherapy +/- bevacizumab.Measurable disease per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group performance status of 0-1
* Must have a life expectancy of at least 12 weeks
* Age > 18 years at time of study entry
* Body weight >30 kg
* Adequate normal organ and marrow function as defined below:

  * Haemoglobin ≥9.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable)
  * Absolute neutrophil count (ANC) > 1.5x10³per mm³
  * Platelet count ≥75x10⁹/L (≥75,000 per mm³)
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
  * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
* If the patient is not in status post hysterectomy, women who are of child-bearing potential willing to use effective methods of contraception including oral contraceptives, intrauterine device, diaphragm with spermicides, and/or abstinence. Women of childbearing potential who have a negative serum pregnancy test and must agree to practice effective birth control throughout their participation in the treatment phase of the study.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
  * Status post hysterectomy
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) 4 weeks prior to the first dose of study drug
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
* Other epithelial tumors (except for adenosquamous carcinoma) defined by WHO histological classification (including neuroendocrine tumors and undifferentiated carcinoma)
* Non-epithelial cervical tumors defined by WHO histological classification: mesenchymal tumors and tumor-like conditions; mixed epithelial and mesenchymal tumors; germ cell tumors; lymphoid and myeloid tumors
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of any investigational products (BVAC-C or durvalumab). The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
* Prior therapy with any anti-PD-1 or anti-PD-L1 inhibitor including durvalumab
* Recurrent/refractory cervical cancer amenable to curative local therapy
* Known severe ischemic heart disease, severe arrythmia and other clinically significant cardiac disease
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-06-14 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Part A : Dose-limiting toxicities(DLTs) | up to 11 weeks
  The primary objective of the part A is to assess the maximum tolerable dose of BVAC-C combined with durvalumab 1500 mg as defined by dose-limiting toxicities (DLTs), and to find the maximum tolerated dose (MTD) that can be safely used for Part B (single arm phase II).
Part B : Evaluate the safety and clinical efficacy, as measured by 6-month PFS rate | 6 Months
  The primary objective of the part B is to evaluate the safety and clinical efficacy, as measured by 6-month PFS rate, of the combination therapy of durvalumab and BVAC-C in patients with HPV 16 or 18 positive cervical cancer recurrent after or refractory to first-line platinum-based chemotherapy +/-bevacizumab.

SECONDARY OUTCOMES:
Best overall response rate(BORR) | 12~24 Months
  • To evaluate the response to the combination therapy as measured by best overall response rate (BORR), 12-month and 24-month disease control rate (DCR), 12-month and-24 month progression free survival (PFS) rate and 12-month and 24-month overall survival (OS) rate.
Disease control rate(DCR) | 12~24 Months
  • To evaluate the response to the combination therapy as measured by best overall response rate (BORR), 12-month and 24-month disease control rate (DCR), 12-month and-24 month progression free survival (PFS) rate and 12-month and 24-month overall survival (OS) rate.
Progression free survival (PFS) rate | 12~24 Months
  • To evaluate the response to the combination therapy as measured by best overall response rate (BORR), 12-month and 24-month disease control rate (DCR), 12-month and-24 month progression free survival (PFS) rate and 12-month and 24-month overall survival (OS) rate.
Overall survival (OS) rate | 12~24 Months
  • To evaluate the response to the combination therapy as measured by best overall response rate (BORR), 12-month and 24-month disease control rate (DCR), 12-month and-24 month progression free survival (PFS) rate and 12-month and 24-month overall survival (OS) rate.
Adverse event(AE) | up to 99 weeks
  • To evaluate the safety of combination therapy of durvalumab and BVAC-C as measured by adverse events (AE), adverse events of special interest (AESI), vital signs, physical examination, safety laboratory tests, including change of lymphocyte subsets from baseline, plasma cytokine level
Adverse events rate of special interest(AESI) | up to 99 weeks
  • To evaluate the safety of combination therapy of durvalumab and BVAC-C as measured by adverse events (AE), adverse events of special interest (AESI), vital signs, physical examination, safety laboratory tests, including change of lymphocyte subsets from baseline, plasma cytokine level

OTHER OUTCOMES:
Programmed death-ligand 1(PD-L1) | 1-2 day
  PD-L1 expression level
Tumor mutational burden(TMB) | 1-2 day
  TBM is a biomarker that can predict the response of PD-L1 to treatment.
Rate of Tumor infiltrating lymphocytes(TIL) | 1-2 day
  Cancers with a DNA repair gene deficiency repair (dMMR) mechanism undergo changes very frequently and accumulate mutations in monomorphic microsatellites (short tandem repeats). And is prone to mismatch errors.
Immune gene expression profile(RNA) | 1-2 day
  We studied immune cell expression profiles for various cancer immune characteristics and confirmed significant differences in OS.
Serum cytokine level(multiplex cytokine assay) | 1-2 day
  Immune cells secrete various cytokines that induce subsequent activation of the immune system. It is worth confirming that BVAC-C can increase blood cytokines.
T cells (ELISPOT) | 1-2 day
  ELISA (The enzyme-linked immunospot) can quantify the cell-mediated immune response with a sensitive technique that can detect cells that produce cytokines at the single cell level. This method of analysis allows for rapid, reproducible, and infrequent direct counting of antigen-specific T cells.
HPV types | 1-2 day
  Biopsy samples will be continuously evaluated to search for biomarkers other than immune profiles and gene signatures that can predict responsiveness to concomitant administration.

IPD SHARING:
Plan to Share IPD: No